CLINICAL TRIAL: NCT05592184
Title: Dual Task During Resistance Training in Patients With Carpal Tunnel Release
Brief Title: Dual Task During Resistance Training in CTR
Acronym: DTRTCTR
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Laura López-Bueno, Clinical Professor, University of Valencia
Other Study IDs: ID0005
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dual task: Exercise (elastic resistance) with dual task The dual task will be self-regulated and will consist of subtracting 3 by 3 from 100, and performing the maximum number of repetitions possible.
  Interventions: Other: Exercise
- Single task: exercise (elastic resistance) without dual task
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The experimental protocol begins with the assessment of self-perceived pain intensity and perceived exertion when using different intensities of elastic resistance, during wrist flexion and extension, at a controlled speed of 1.5sec/ phase. To assess the intensity at which they will work, participants will perform 2 repetitions and will be allowed a rest of 60s between sets until they obtain a score of 3 on the Borg CR10 scale. Exercises should be performed with the subject's available ROM. Participants are asked to move their body and trunk as little as possible and to perform the exercise smoothly, without stopping or accelerating. The exercise will be performed in a seated position, with the back supported by the backrest and the forearm resting on a table, with the shoulders and elbows bent at 90o, leaving the wrist free, with the elastic bands held under the feet (stepping on them).

SUMMARY:
Carpal tunnel syndrome (CTS) is a highly prevalent peripheral compressive neuropathy of the upper extremity. CTS is characterised by the presence of pain, tingling sensations and paraesthesia in the median nerve territory. Symptom severity and pain are commonly modulated by psychosocial factors (e.g. catastrophic thinking and kinesiophobia).

The objective of this study will be (1) to evaluate the effect of dual-task on the maximum number of repetitions possible and pain during rubber band training in patients with carpal tunnel syndrome undergoing surgery; (2) to determine the influence of psychosocial factors on the response to dual-task exercise.

Patients will voluntarily participate in the study, which will be conducted at the Hospital Clínico Universitario de Valencia, during the months of November 2022 to December 2022. All participants will be informed of the aims and content of the research and written informed consent will be obtained. The study will conform to the Declaration of Helsinki and will be approved by the local ethics committee.

The experimental protocol begins with the assessment of self-perceived pain intensity and perceived exertion when using different intensities of elastic resistance, during wrist flexion and extension, at a controlled speed of 1.5sec/ phase. To assess the intensity at which they will work, participants will perform 2 repetitions and will be allowed a rest of 60s between sets until they obtain a score of 3 on the Borg CR10 scale. For this purpose, 1.5 m long elastic bands, pre-stretched to approximately 25% of their initial length, in yellow, red, green, blue, black, silver and gold (TheraBand CLX, The Hygenic Corporation, Akron, OH, USA), will be progressively used starting from the lowest available elastic resistance (i.e. yellow). This intensity is selected because it appears to correspond to a resistance equivalent to 30% of 1RM and is considered a light intensity. Exercises should be performed with the subject's available ROM. Participants are asked to move their body and trunk as little as possible and to perform the exercise smoothly, without stopping or accelerating. The exercise will be performed in a seated position, with the back supported by the backrest and the forearm resting on a table, with the shoulders and elbows bent at 90 grades, leaving the wrist free, with the elastic bands held under the feet (stepping on them).

During the week of familiarisation and analysis of acute effects, subjects will attend 2 sessions, separated by 2 rest days in between, where they will perform 2 conditions/session (4 conditions in total at the end of the study), in a counterbalanced manner, with 10 minutes rest between each condition: 1) perform the highest number of wrist flexion repetitions with the appropriate resistance; 2) perform the highest number of wrist flexion repetitions with the appropriate band, and following a dual task; 3) perform the highest number of wrist extension repetitions with the appropriate band; 4) perform the highest number of wrist extension repetitions with the appropriate band, and following a dual task.

The dual task will be self-regulated and will consist of subtracting 3 by 3 from 100, and performing the maximum number of repetitions possible. The subject will perform the mathematical operation aloud, without being corrected, but if they get stuck on a number or operation, they will have to be told to continue subtracting from that number or from another, so that they do not stop performing the operations. At the end of each condition, the subject will be asked about the perceived difficulty of the self-regulated mathematical task (where 0 is not difficult at all and 10 is the maximum difficulty), and the maximum number of repetitions performed will be recorded. The pressure points and VAS will then be measured again.

After the familiarisation week and the analysis of acute effects, subjects will be randomly distributed into two conditions: 1) exercise with dual task; 2) exercise without dual task. The exercises performed will be the same as during the familiarisation week, as well as the guidelines for performing them. Each condition shall be evaluated with a time-out (Crossover design).

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of CTS according to international clinical guidelines
* Patients referred for rehabilitation after carpal tunnel release surgery
* Agree to participate

Exclusion Criteria:

* Inability to understand instructions.
* Uncontrolled mental health pathology.
* Cognitive problems.
* Previous surgery on the upper extremity. • Complex regional pain syndrome

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men and women aged 20-60 years with a medical diagnosis of CTS according to international clinical guidelines will be candidates for the present study. Patients receiving rehabilitation following carpal tunnel release surgery will be potentially eligible
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Maximum number of repetitions possible | 1 day
  The maximum number of repetitions possible in each of the conditions shall be counted (BORG 3/10)
Pain intensity | 2 days
  The VAS is a 100 millimeter (mm) line used to assess self-perceived pain intensity in research. At the left end of the line is a small text indicating "no pain" and at the right end of the line is a small text stating "maximum bearable pain". The patient marks a point on the scale and then the clinician or researcher quantifies the number of mm marked by the patient. Thus, the range of self-perceived pain intensity travels from 0-100 mm.

SECONDARY OUTCOMES:
Kinesiophobia | 1 day
  Kinesiophobia will be assessed using the Spanish version of the Tampa Kinesiophobia Scale in a self-recorded manner. This instrument has shown adequate reliability (showing an internal consistency of α=0.79). The total score ranges from 11 to 44 points, with higher levels of kinesiophobia occurring the higher the score on the scale [17]. In addition, kinesiophobia specific to the type of exercise performed will be assessed, with a self-perceived scale from 0 to 10, where patients will indicate the fear of performing all possible repetitions during a strength exercise.
Catastrophizing | 1 day
  The level of Catastrophism will be assessed through the self-recorded Pain Catastrophism Scale, which consists of 13 items describing different thoughts and feelings associated with pain. The scale has 5 grades, being 0 not at all, 1 a little, 2 moderately, 3 a lot and 4 all the time. The subject has to mark his or her situation in each case. The scale consists of 13 items in total (0-52 points). Higher scores indicate higher levels of pain catastrophism. This questionnaire has a minimum detectable change of 10.45 points and has shown excellent psychometric reliability data (α=0.94). The cut-off point for early detection of people with a tendency towards pain catastrophizing is 11 points.
Self-efficacy | 1 day
  The Perceived Chronic Pain Self-Efficacy questionnaire contains 19 items and assesses 3 domains with good psychometric reliability values: self-efficacy for pain management (α=0.72), physical functioning (α=0.98) and symptom management (α=0.85). Each item is scored from 0-10, with 0 being "not at all able" and 10 being "fully able". The main objective of this questionnaire is to assess the perceived self-efficacy and ability to cope with the consequences of pain in patients with chronic pain. Furthermore, this questionnaire has a criterion (concurrent) validity value of r=0.75.
Pressure Pain Thresholds | 2 days (baseline and post exercise)
  The Algometer (Wagner Instruments, Greenwich, CT, USA), will be used in this study. It consists of a round rubber disc (1 cm2 surface area) attached to a pressure (force) gauge. The gauge displays values in kilograms, but as the surface area of the rubber tip is 1 cm2, the readings are expressed in kg/cm2. The range of values of the pressure algometer is from 0 to 10 kg, in 0.1 kg intervals. Pressure is applied at a rate of 0.31 kg/s or 1 kg every 3 seconds. Previous studies have reported that the intra-examiner reliability of this procedure ranges between 0.6 and 0.97, while the inter- examiner reliability ranges between 0.4 and 0.98. Pressure pain thresholds will be carried out bilaterally (affected and unaffected side) on the carpal tunnel (distal to the scar) and lateral epicondyle on the unaffected limb.This variable will be measured pre and immediate post-exercise
The Symptom Severity Questionnaire | 1 day
  The Symptom Severity Questionnaire consists of 11 questions, each offering 5 response options, from 1 (no symptoms) to 5 (most severe/frequent). The score for each subscale is weighted to obtain an average ranging from 1 to 5 points. This questionnaire will be administered pre- and post-intervention.
The Functionality Questionnaire | 1 day
  The Functionality Questionnaire includes 8 questions assessing difficulty in performing everyday tasks (opening a new or very tight bottle, writing, turning a key, preparing food, etc.). The score for each subscale is weighted to obtain an average ranging from 1 to 5 points. This questionnaire will be administered pre- and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain